CLINICAL TRIAL: NCT01251939
Title: Observational Study of Near Infrared Spectroscopy to Monitor Renal and Splanchnic Oxygenation During Ibuprofen Treatment for Patent Ductus Arterious in Preterm Infants
Brief Title: Changes in Renal and Splanchnic Oxygenation During Ibuprofen Treatment for Patent Ductus Arterious
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Nilufer Guzoglu, MD, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: n7860088
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Ductus Arteriosus, Patent
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment with ibuprofen: Gestational age <32 weeks and <1500 g, postnatal age older than 48 hours and echocardiographic evidence of hemodynamically significant PDA
  Interventions: Device: Near-infrared spectroscopy (NIRS)
- Controls: Gestational age <32 weeks and <1500 g, postnatal age older than 48 hours and without significant PDA
  Interventions: Device: Near-infrared spectroscopy (NIRS)

INTERVENTIONS:
Device: Near-infrared spectroscopy (NIRS) — Non-invasive monitoring device measures the quantity of reflected light photons as a function of two wavelengths, and determines the spectral absorption of the underlying tissue.
  Other Names: INVOS 4100 oximeter, Somanetics,

SUMMARY:
Patent ductus arterious(PDA)is frequently seen and potentially pathologic in preterm infants. Near-infrared spectroscopy is a simple bedside tool to analyse the changes in the renal and splanchnic tissue oxygenation index and fractional tissue oxygen extraction and may be helpful to measure effects of ibuprofen treatment for PDA in preterm infants.

DETAILED DESCRIPTION:
Patent ductus arterious (PDA) is the most common cardiovascular abnormality in preterm infants.There are clear associations between a PDA and decreased renal and splanchnic blood flow. The aim is to monitor, using near-infrared spectroscopy, the effect of ibuprofen on the fractional tissue (renal and mesenteric) oxygen extraction (FTOE) in preterm newborns during ibuprofen of the treatment PDA.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 weeks and <1500 g
* Echocardiographic evidence of hemodynamically significant patent ductus arterious

Exclusion Criteria:

* Major congenital anomalies
* Intraventricular hemorrhage of grade 3 within the previous 24 hours
* Serum creatinine level 1.5 mg%,serum urea nitrogen concentration >50 mg%,
* Platelet count 60 000/mL3, a tendency to bleed (defined by the presence of hematuria, blood in the endotracheal aspirate, gastric aspirate, or stools and/or oozing from puncture sites)
* Hyperbilirubinemia necessitating exchange transfusion

Min Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants who born in Zekai Tahir Burak Maternity and Teaching Hospital between january 2011 and january 2012 and met the entry criteria first underwent echocardiography and cranial ultrasonography.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilufer Guzoglu, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity and Teaching Hospital, Ankara, Turkey (Türkiye)